CLINICAL TRIAL: NCT04097054
Title: The 3P Trial: Preoperative Planning and Preparation of Complex and Rare Procedures in GI Surgery: Can we Improve the Operative Workflow and Patient Outcomes?
Brief Title: The 3P Trial: Preoperative Planning and Preparation of Complex and Rare Procedures in GI Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3P2019
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Surgical Procedures, Operative
Keywords: operative procedures; intraoperative monitoring; budgetary control

STUDY DESIGN:
Intervention Model Description: A single centre randomized open label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the interventional arm are operated after augmented planning of the procedure. The plan is prepared by the surgeon and made available to the study team a day prior to the procedure and on a screen in the OR during the procedure. The plan includes the current and next operative step, the used equipment and the approximate time used as well as the estimated time of when the procedure will end.
  Interventions: Procedure: Augmented preoperative planning
- Control (No Intervention): In the control cases no particular planning and distribution of operative plan is performed. The standard preparation only includes the distribution of information on the desired positioning of the patient, necessary special equipment and the overall estimated OR time.

INTERVENTIONS:
Procedure: Augmented preoperative planning — The study investigates the impact of augmented preoperative planning on OR time variance in complex and rare visceral surgical procedures.
  Arms: Intervention

SUMMARY:
The aim of the present study is to develop, implement a planning tool for rare and complex visceral surgical procedures. With the successful implementation of the planning tool the study will contribute to the improvement of intraoperative processes and their outcome in low volume surgery and offer an alternative to continued centralization of surgical care especially in case of geographical or disease specific premises.

DETAILED DESCRIPTION:
The quality of the intraoperative process is still a blind spot, when it comes to clinical surgical research in the operating room. In contrast to pre and postop process optimization with tools like the World Health Organization (WHO) checklist or the Enhanced Recovery after Surgery (ERAS) protocol intraoperative processes tend to be poorly defined especially in rare and complex visceral surgery (e.g. esophageal, pancreatic rectal resection, sarcoma surgery, revisional bariatric surgery). This leads to delay, increased stress of the operating team and increased intraoperative mistakes and eventually increased complication rates. From previous investigations we know that step by step planning and briefing of the entire OR Team can reduce operative interruptions. With the development of a dedicated planning tool which allows to create and distribute step by step protocols for rare and complex visceral surgical procedures to the entire OR Team we hope to decrease delays and reduce OR time variance.

Objective: Development and implementation of a planning tool for rare and complex visceral surgical procedures.

Outcomes: Primary outcome: (delay/variability) operative times as defined as time from skin incision to skin closure

Secondary outcomes:

* Costs
* Influence of preoperative augmented planning on degree of and quality of teaching
* Level of stress of each operating team member
* Number of intraoperative mistakes
* Number and severity of intraoperative and postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older,
* indication for a complex and rarely performed visceral surgical procedure (e.g. esophagectomy, Whipple operation, Gastrectomy, complex hepatobiliary surgery, multivisceral resections, rectal cancer surgery, revisional bariatric surgery),
* patient's written informed consent
* consent of the involved operating team

Exclusion Criteria:

* age younger than 18 years,
* Emergency surgery or a time from outpatient visit to the operation <8 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
delay/variability of operative time | 1 year, measured after every operation
  The primary outcome is the (delay/variability) of operative time as defined as time from skin incision to skin closure that will be recorded with the hospital OR planning program (Ismed Protect Data) and compared to preoperatively planned times.

SECONDARY OUTCOMES:
Costs | 1 year, calculated after every case once patient is dismissed
  Costs will be calculated as intraoperative delay compared to preoperative planning in minutes multiplied with the OR minute costs of the institution in addition to the average salaries per minute of the involved surgical staff. OR minute costs will be calculated by dividing the OR and anesthesia cost units through the overall operative time in the institution. The OR cost unit includes the personnel expenses for operating nurses and other staff (including cleaner and others) as well as maintenance costs (single use equipment, depreciation on buildings and running expenses like water and electricity etc. The cost unit anesthesia includes all expenses for personnel (doctors and nurses), depreciation for respirators and other devices as well as expandable materials.
Level of stress | 1 year, measured during every operation
  Level of stress of each operating team member will be assessed directly postoperatively with a Visual Analogue Scale (VAS) report (operated on an ipad for data collection). The VAS Scale will consist of a 0 (no stress) to 7 (maximum stress) item scale.
Number of intraoperative mistakes | 1 year, measured during every operation and compiled after the operation is finished
  Number of intraoperative mistakes will be recorded with a pedal button operated by the first assistant on the demand of the lead surgeon.
Number and severity of intraoperative complications | 1 year, measured during every operation and compiled after the operation
  Number and severity of intraoperative complications will be assessed directly postoperatively by the lead surgeon and or first assistant, audio video records are available for review purposes. Postoperative complications will be recorded after discharge on the basis of discharge summary and proceeding notes of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Marco von Strauss und Torney, PD Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel/Dep. of General and Visceral Surgery, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No